CLINICAL TRIAL: NCT01269372
Title: Evaluation of Capsule Endoscopy With PillCam® Colon 2 in Visualization of the Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Device Feasibility
Other Study IDs: MA-203
Record Dates: First submitted 2010-11-18; First posted 2011-01-04 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Lesions
Keywords: polyps; capsule endoscopy; colonoscopy
MeSH Terms: conditions — Polyps | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- PillCam Colon 2 and Standard Colonoscopy (Other): All subjects received Capsule Endoscopy (CE) using the PillCam Colon 2 followed by a standard colonoscopy.
  Interventions: Device: PillCam Colon 2; Device: Colonoscopy

INTERVENTIONS:
Device: PillCam Colon 2 — Each subject will be required to follow a bowel preparation regimen and will undergo Capsule Endoscopy (CE).
  Following capsule ingestion and depending on capsule progression through the digestive tract subjects will be required to take an additional volume of laxatives in order to enhance capsule propulsion and maintain adequate cleansing of the colon.
Device: Colonoscopy — The colonoscopy procedure will be scheduled approximately 4-6 weeks after the CE procedure, and the colonoscopy bowel preparation will be the same as the bowel preparation for CE.

SUMMARY:
This pilot, multi center study will establish the effectiveness of Given PillCam® Platform with the PillCam® Colon 2 Capsule as demonstrated by the identification of subjects with polyps, compared to standard colonoscopy.

This study will also use to evaluate the administrative feasibility and data management of study design.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 50 - 75 years of age, and an appropriate candidate for polyp screening.
2. Subject received an explanation about the nature of the study and agrees to provide written informed consent.

Exclusion Criteria:

1. Subject has a history of colorectal cancer
2. Subjects with history of any positive colon assessment (including CT, colonoscopy, sigmoidoscopy etc.),
3. Subject with history of negative colon assessment (including CT, colonoscopy, sigmoidoscopy etc.) < 5 years.
4. Subject has a first degree relative diagnosed with colorectal cancer before the age of 60 years old or 2 (or more) first degree relatives diagnosed with colorectal cancer at any age.
5. Subject is suspected or diagnosed with familial adenomatous polyposis.
6. Subject is suspected or diagnosed with hereditary nonpolyposis colon cancer.
7. Subject is suspected or diagnosed with inflammatory bowel disease, or chronic ulcerative colitis or Crohn's disease.
8. Subject is suspected or diagnosed with hematochezia, melena, Fe deficiency anemia or any other rectal bleeding., including positive FOBT test of any variety
9. Subject is suspected or diagnosed with bowel obstruction.
10. Subject has dysphagia or any swallowing disorder.
11. Subject has congestive heart failure.
12. Subject has Diabetes.
13. Subject has had prior abdominal surgery of the gastrointestinal tract in the last 6 months or other uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
14. Subject has a cardiac pacemaker or other implanted electro medical device.
15. Subject has any allergy or other known contraindication to the medications used in the study.
16. Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
17. Subject with any condition believed to have an increased risk for capsule retention such as intestinal tumors, radiation enteritis, and incomplete colonoscopies due to obstructions or NSAID enteropathy.
18. Subject with strictures, fistulas and/or chronic constipation.
19. Subject with history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters.
20. Subject with known gastrointestinal motility disorders.
21. Subject has known delayed gastric emptying.
22. Subject has any condition, which precludes compliance with study and/or device instructions.
23. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
24. Subject suffers from life threatening conditions.
25. Subject currently participating in another clinical study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, Prof., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Gastroenterology Associates of Tidewater, Chesapeake, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Reporting Group: This was a single center study where 30 patients were enrolled. No formal sample sizing has been performed as this study was a pilot for a larger multicenter trial.
  All subjects that were enrolled in this study were indicated and scheduled to undergo colonoscopy based on their age and demographics for screening for polyps.
Period: Overall Study
Arm/Group | Reporting Group
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reporting Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 52.57 [50 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 30
Thirty patients were enrolled in the study. [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of the PillCam® Colon 2 Capsule Endoscopy (CE) for Polyps Per Subject - Sensitivity
Description: PillCam® Colon 2 Capsule Endoscopy (CE) compared to standard colonoscopy in detecting subjects with polyps equal to or larger than 6 mm and 10 mm as measured by Sensitivity. A positive event was defined as per optical colonoscopy polyp size measurement. Standard colonoscopy is the gold standard.
Time Frame: Up to 6 weeks
Population: The accuracy parameters were calculated per subject analysis, i.e. the accuracy events were generated by the larger polyp identified in a given subject.
Measure: Number (95% Confidence Interval); unit: percentage of sensitivity
Groups:
- PillCam® Colon 2 Followed by Standard Colonoscopy - >6mm Polyp: All subjects received PillCam Colon 2 followed by standard colonoscopy 4-6 week after CE procedure. Sensitivity is presented for the detection of subjects with polyp >= 6mm
- PillCam® Colon 2 Followed by Standard Colonoscopy 10mm Polyp: All subjects received PillCam Colon 2 followed by standard colonoscopy 4-6 week after CE procedure. Sensitivity is presented for the detection of subjects with polyp >= 10mm
Arm/Group | PillCam® Colon 2 Followed by Standard Colonoscopy - >6mm Polyp | PillCam® Colon 2 Followed by Standard Colonoscopy 10mm Polyp
Number analyzed (Participants) | 30 | 30
percentage of sensitivity | 83 [42 to 99] | 50 [9 to 91]

2. Primary Outcome: Accuracy of the PillCam® Colon 2 Capsule Endoscopy (CE) for Polyps Per Subject - Specificity
Description: PillCam® Colon 2 Capsule Endoscopy (CE) compared to standard colonoscopy in detecting subjects with polyps equal to or larger than 6 mm and 10 mm as measured by Specificity. A positive event was defined as per optical colonoscopy polyp size measurement. Standard colonoscopy is the gold standard.
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of specificity
Arm/Group | PillCam® Colon 2 Followed by Standard Colonoscopy - >6mm Polyp | PillCam® Colon 2 Followed by Standard Colonoscopy 10mm Polyp
Number analyzed (Participants) | 30 | 30
percentage of specificity | 92 [73 to 99] | 100 [86 to 100]

3. Secondary Outcome: Accuracy of the PillCam® Colon 2 Capsule Endoscopy (CE) Detecting Polyps Per Location - Sensitivity
Description: PillCam® Colon 2 Capsule Endoscopy (CE) compared to standard colonoscopy was evaluated by clustered sensitivity for polyps equal to or larger than 6 mm and 10 mm as measured by Sensitivity. A positive event was defined as per optical colonoscopy polyp size measurement. Standard colonoscopy is the gold standard.
Time Frame: Up to 6 weeks
Population: The accuracy parameters were calculated per segment analysis, i.e. the accuracy events were generated by the larger polyp identified in a given location (5 segments).
Measure: Number (95% Confidence Interval); unit: percentage of sensitivity
Groups:
- PillCam® Colon 2 Followed by Standard Colonoscopy - >6mm Polyp: All subjects received PillCam Colon 2 followed by standard colonoscopy 4-6 week after CE procedure. Sensitivity is presented for the detection of polyps >= 6mm per segment
- PillCam® Colon 2 Followed by Standard Colonoscopy 10mm Polyp: All subjects received PillCam Colon 2 followed by standard colonoscopy 4-6 week after CE procedure. Sensitivity is presented for the detection for polyp >= 10mm per segment
Arm/Group | PillCam® Colon 2 Followed by Standard Colonoscopy - >6mm Polyp | PillCam® Colon 2 Followed by Standard Colonoscopy 10mm Polyp
Number analyzed (Participants) | 30 | 30
percentage of sensitivity | 80 [48 to 95] | 33 [6 to 80]

4. Secondary Outcome: Accuracy of the PillCam® Colon 2 Capsule Endoscopy (CE) Detecting Polyps Per Location - Specificity
Description: PillCam® Colon 2 Capsule Endoscopy (CE) compared to standard colonoscopy was evaluated by clustered sensitivity for polyps equal to or larger than 6 mm and 10 mm as measured by Specificity. A positive event was defined as per optical colonoscopy polyp size measurement. Standard colonoscopy is the gold standard.
Time Frame: Up to 6 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of specificity
Groups:
- PillCam® Colon 2 Followed by Standard Colonoscopy - >6mm Polyp: All subjects received PillCam Colon 2 followed by standard colonoscopy 4-6 week after CE procedure. Specificity is presented for the detection of polyps >= 6mm per segment
- PillCam® Colon 2 Followed by Standard Colonoscopy 10mm Polyp: All subjects received PillCam Colon 2 followed by standard colonoscopy 4-6 week after CE procedure. Specificity is presented for the detection for polyp >= 10mm per segment
Arm/Group | PillCam® Colon 2 Followed by Standard Colonoscopy - >6mm Polyp | PillCam® Colon 2 Followed by Standard Colonoscopy 10mm Polyp
Number analyzed (Participants) | 30 | 30
percentage of specificity | 96 [92 to 99] | 100 [97 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events were collected and documented until the end of Colonoscopy procedure, which was scheduled 4-6 weeks after the PillCam Colon 2 CE procedure and was the end of the study.
Arm/Group | PillCam Colon 2 and Standard Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 6/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PillCam Colon 2 and Standard Colonoscopy (N=30)
alergic reaction to adhesive (Skin and subcutaneous tissue disorders) | 2 (2) — Related to capsule procedure
Globus Hystericus (Gastrointestinal disorders) | 1 (1) — Related to capsule procedure
abdominal pain (General disorders) | 2 (2) — Related to colon prep
diarrhea (Gastrointestinal disorders) | 1 (1) — Related to colon prep
nausea (Gastrointestinal disorders) | 1 (2) — Related to colon prep
headache (Gastrointestinal disorders) | 1 (1) — Related to prep
vomiting (Gastrointestinal disorders) | 1 (1) — Related to colon prep

LIMITATIONS AND CAVEATS:
This was a feasibility study, in accordance with the definition of a feasibility study within the ACT checklist. The feasibility study was used as preparation to study pivotal study number MA- 204 NCT01372878 which has results posted on CT.gov.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No